CLINICAL TRIAL: NCT03988023
Title: A Randomized, Controlled, Double-Blind Study to Evaluate the Efficacy and Safety of an Intra-Articular Injection of Ampion in Adults With Pain Due to Severe Osteoarthritis of the Knee.
Brief Title: Study of Ampion for the Treatment of Pain and Function in Patients With Severe Osteoarthritis of the Knee.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The AP-013 study was prematurely terminated by the sponsor after Data Safety Monitoring Board (DSMB) guidance.
Sponsor: Ampio Pharmaceuticals. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP-013
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Results first posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-08

CONDITIONS: Severe Osteoarthritis of the Knee
Keywords: Osteoarthritis; osteoarthritis of the knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — aspartyl-alanyl-diketopiperazine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMPION™ 4 mL dose (Experimental): 4 mL injection of Ampion
  Interventions: Biological: Ampion
- Saline (Placebo Comparator): 4 mL injection of placebo
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: Ampion — 4 mL injection of Ampion
  Arms: AMPION™ 4 mL dose
Drug: Saline — Saline solution, 4 mL, single intra-articular injection
  Other Names: 0.9% Saline
  Arms: Saline

SUMMARY:
The purpose of this study is to confirm the safety and efficacy of Ampion for the treatment of pain and function in patients with severe osteoarthritis of the knee.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, single dose design.

The co-primary trial objectives are to evaluate the greater efficacy for pain improvement and function improvement of 4 mL Ampion versus saline intra-articular (IA) injection when applied to patients suffering from severe osteoarthritis of the knee (OAK). Efficacy will primarily be assessed with WOMAC A pain and WOMAC C function scores.

Mean change in the WOMAC A weekly pain scores from Baseline to Week 12 will be compared between Ampion and saline control. Mean change in WOMAC C function score will be compared between Ampion and saline control. This will test whether Ampion is superior to saline in improving pain and function.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent to participate in the study
* Willing and able to comply with all study requirements and instructions of the site study staff
* Must be ambulatory
* Index knee must be symptomatic for greater than 6 months with a clinical diagnosis of OAK and supported by radiological evidence (Kellgren-Lawrence Grade 4) that is not older than 6 months prior to the date of screening
* Moderate to moderately-severe osteoarthritis (OA) pain in the index knee (rating of at least 1.5 on the WOMAC Index 3.1 as measured by 5-point Likert Pain Subscale) assessed at screening
* Ability to temporarily discontinue nonsteroidal anti-inflammatory drug (NSAID) for 48 hours prior to scheduled clinical efficacy evaluations
* No analgesia (including acetaminophen [paracetamol]) taken 12 hours prior to an efficacy measure
* No known clinically significant liver abnormality (e.g. cirrhosis, transplant, etc.).

Exclusion Criteria:

* As a result of medical review and screening investigation, the Principal Investigator considers the patient unfit for the study
* A history of allergic reactions to human albumin (reaction to non-human albumin such as egg albumin is not an exclusion criterion)
* A history of allergic reactions to excipients in 5% human albumin (N-acetyltryptophan, sodium caprylate)
* Presence of tense effusions
* Inflammatory or crystal arthropathies, acute fractures, history of aseptic necrosis or joint replacement in the affected knee, as assessed locally by the Principal Investigator
* Isolated patella femoral syndrome, also known as chondromalacia
* Any other disease or condition interfering with the free use and evaluation of the index knee for the duration of the trial (e.g. cancer, congenital defects, spine osteoarthritis)
* Major injury to the index knee within the 12 months prior to screening
* Severe hip osteoarthritis ipsilateral to the index knee
* Any pain that could interfere with the assessment of index knee pain (e.g. pain in any other part of the lower extremities, pain radiating to the knee)
* Any pharmacological or non-pharmacological treatment targeting OA started or changed during the 4 weeks prior to randomization or likely to be changed during the duration of the study
* Use of the following medications:

  1. No IA injected pain medications in the study knee during the study
  2. No analgesics containing opioids. NSAIDs may be continued at levels preceding the study, however may not be used 48 hours prior to efficacy evaluations, and acetaminophen is available as a rescue medication during the study from the provided supply
  3. No topical treatment on osteoarthritis index knee during the study
  4. No significant anticoagulant therapy (e.g. Heparin or Lovenox) during the study (treatment such as Aspirin and Plavix are allowed)
  5. No systemic treatments that may interfere with safety or efficacy assessments during the study
  6. No immunosuppressants
  7. No use of corticosteroids > 10 mg prednisolone equivalent per day
  8. If corticosteroid use is ≤ 10 mg prednisolone equivalent per day, and if clinically indicated, subjects should be allowed to decrease their corticosteroid use. Additionally, some subjects may need to increase their steroid dose to treat worsened symptoms in the treated knee, and subjects who increase their corticosteroid dose above their starting dose of corticosteroid during the study will be treated as "treatment failures" for efficacy analysis
* No human albumin treatment in the 3 months before randomization or throughout the duration of the study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1043 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Levy, M.D., Study Director — Ampio Pharmaceuticals. Inc.
Locations (1):
- Denver Metro Orthopedics, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of subjects occurred in medical clinics from June 2019 to March 2020.
Pre-assignment Details: No pharmacological or non-pharmacological treatment targeting osteoarthritis (OA) started or changed during the 4 weeks prior to randomization or likely to be changed during the duration of the study.
Groups:
- Ampion 4 mL Dose: 4 mL Injection of Ampion
- Placebo 4 mL Dose: 4 mL Injection of Placebo
Period: Overall Study
Arm/Group | Ampion 4 mL Dose | Placebo 4 mL Dose
Started | 520 | 523
Completed | 235 | 235
Not Completed | 285 | 288
Not completed — Non-compliance | 3 | 0
Not completed — Withdrawal by Subject | 39 | 37
Not completed — Adverse Event | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 5 | 8
Not completed — Sponsor decision to terminate follow up | 10 | 12
Not completed — Lack of Efficacy | 3 | 1
Not completed — COVID-19 pandemic | 225 | 227

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ampion 4 mL Dose | Placebo 4 mL Dose | Total
Number analyzed (Participants) | 520 | 523 | 1043
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9.2) | 64.7 (9.2) | 64.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304 | 342 | 646
  Male | 216 | 181 | 397
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 23 | 51
  Not Hispanic or Latino | 491 | 495 | 986
  Unknown or Not Reported | 1 | 5 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 98 | 83 | 181
  White | 410 | 429 | 839
  More than one race | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 520 | 523 | 1043
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.8 (8.1) | 34.7 (8.5) | 34.3 (8.3)
WOMAC Pain [Mean (Standard Deviation); unit: Score on a scale] — The Western Ontario and McMaster Universities Arthritis Index (WOMAC) 3.1 evaluates Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright.
  Subjects respond to each subscale by using a 5-point Likert score. (0=none; 1=mild; 2=moderate; 3=severe; 4=extreme). Mean of the 5 scores constitutes the Baseline Pain Score.
  The minimum score on this scale is 0, and the maximum score is 4. Higher scores are indicative of higher levels of self-reported pain.
  Score on a scale | 2.34 (0.69) | 2.40 (0.70) | 2.37 (.69)
WOMAC Function [Mean (Standard Deviation); unit: Score on a scale] — WOMAC 3.1 evaluates Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in/out of a car, shopping, putting on/taking off socks, rising from bed, lying in bed, getting in/out of bath, sitting, getting on/off toilet, heavy/light domestic duties.
  Subjects respond to each by using a 5-point Likert score. (0=none; 1=mild; 2=moderate; 3=severe; 4=extreme).
  Mean of the 17 scores constitutes the Baseline Function Score. Minimum score is 0; maximum is 4. Higher scores indicate of higher levels of limitations of self-reported physical function.
  Score on a scale | 2.43 (0.70) | 2.45 (0.72) | 2.44 (0.71)

OUTCOME MEASURES:

1. Primary Outcome: Change in Knee Pain
Description: Mean Change in WOMAC A Pain (Western Ontario and McMaster Universities Arthritis Index) score from Baseline to 12 weeks. 5-point Likert scale (0=none to 4=extreme). A negative difference constitutes a decrease in pain with a greater negative value indicating a greater reduction in pain.
Time Frame: Scored at Baseline and 12 Week
Population: Intent to Treat (ITT)
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Ampion 4 mL Dose | Placebo 4 mL Dose
Number analyzed (Participants) | 520 | 523
Score on a scale | -0.66 [-0.73 to -0.61] | -0.71 [-0.76 to -0.64]
Statistical Analysis 1: Comparison: Ampion 4 mL Dose vs Placebo 4 mL Dose; Test type: Superiority; p = 0.32, MMRM

2. Primary Outcome: Change in Knee Function
Description: Mean change in WOMAC C function score (Western Ontario and McMaster Universities Arthritis Index) from Baseline to 12 weeks. 5-point Likert scale indicating limitation of function (0=none to 4=extreme). A greater negative value indicates a improvement in function.
Time Frame: Scored at Baseline and 12 weeks.
Population: Intent to Treat (ITT)
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Ampion 4 mL Dose | Placebo 4 mL Dose
Number analyzed (Participants) | 520 | 523
Score on a scale | -0.68 [-0.75 to -0.62] | -0.73 [-0.79 to -0.67]
Statistical Analysis 1: Comparison: Ampion 4 mL Dose vs Placebo 4 mL Dose; Test type: Superiority; p = 0.30, MMRM

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Patients will be followed for the occurrence of Adverse Events (AEs) until 24 weeks after the first dose of study medication.
Arm/Group | Ampion 4 mL Dose | Placebo 4 mL Dose
All-Cause Mortality (participants affected / at risk) | 1/520 | 0/523
Serious Adverse Events (participants affected / at risk) | 16/520 | 11/523
Other Adverse Events (participants affected / at risk) | 154/520 | 162/523
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ampion 4 mL Dose (N=520) | Placebo 4 mL Dose (N=523)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (2)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Device breakage (Product Issues) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ampion 4 mL Dose (N=520) | Placebo 4 mL Dose (N=523)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (33) | 35 (41)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 6 (6)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 8 (8) | 7 (8)
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Dizziness (Nervous system disorders) | 1 (1) | 6 (6)
Headache (Nervous system disorders) | 5 (5) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (4)
Hypertension (Vascular disorders) | 7 (7) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (5)
Injection site pain (General disorders) | 5 (5) | 2 (2)
Influenza (Infections and infestations) | 2 (2) | 6 (6)
Nasopharyngitis (Infections and infestations) | 12 (12) | 12 (12)
Sinusitis (Infections and infestations) | 18 (19) | 15 (18)
Upper respiratory tract infection (Infections and infestations) | 14 (14) | 11 (11)
Urinary tract infection (Infections and infestations) | 8 (8) | 11 (11)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 6 (6)
Bronchitis (Infections and infestations) | 6 (6) | 4 (4)
Sciatica (Nervous system disorders) | 2 (2) | 5 (5)

LIMITATIONS AND CAVEATS:
The AP-013 study was prematurely terminated by the sponsor after Data Safety Monitoring Board (DSMB) guidance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT03988023/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT03988023/SAP_001.pdf